CLINICAL TRIAL: NCT06100068
Title: Hyperventilation and Oxygenation to Increase Breath Hold in Breast Cancer Irradiation Treatment (HOBBIT) 3: Mental Exercises and Temporal Alteration
Brief Title: HOBBIT 3: Mental Exercises and Temporal Alteration
Acronym: HOBBIT-META
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: EC/2023/0256 (PA-2023-0017)
Record Dates: First submitted 2023-10-03; First posted 2023-10-25 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Breast Neoplasm; Radiotherapy; Breath Holding; Mental Test
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard L-DIBH (Active Comparator): Starts with 2 sessions of normal L-DIBH followed by 2 sessions of L-DIBH combined with mental exercises.
  Interventions: Behavioral: Mental Exercises and Temporal Alteration
- Intervention L-DIBH (Experimental): Starts with 2 sessions of of L-DIBH combined with mental exercises followed by 2 sessions of normal L-DIBH.
  Interventions: Behavioral: Mental Exercises and Temporal Alteration

INTERVENTIONS:
Behavioral: Mental Exercises and Temporal Alteration — Mental exercises during L-DIBH to distort the awareness of passage of time

SUMMARY:
In the HOBBIT-trial by Vakaet et al. A protocol was developed to increase breath-hold time using (voluntary) hyperventilation and oxygenation to achieve DIBH times around 3 minutes.

Multiple non-medical interventions are being investigated to prolong a L-DIBH that are feasible in clinical practice. One of these methods will be to alter the time perception of the subjects. It has been noted in multiple studies (both medical and not) that slowing a person's perception of time results in an increase in breath-hold time. This alteration in time perception can be achieved with the use of a slowed clock as well as the usage of mental or physical exercises to preoccupy the subjects.

Volunteers will then be randomised into either the standard arm or the intervention arm. The intervention arm will follow standard protocol regarding DIBH preparation, though during the L-DIBH they will be asked to perform a simple mental exercise on a tablet. After 2 sessions of 3 L-DIBHs each, there will be a cross-over to the other arm in order to ascertain comfort and preference with each technique.

DETAILED DESCRIPTION:
Adjuvant radiation therapy has a well-established role in the treatment of breast cancer complementing surgery and systemic treatment, improving survival and local control in both local and regional disease. The long-term follow-up, however, does show increased cardiac morbidity and mortality. The risk of heart disease is greatest in patients receiving a higher heart dosage i.e., left sided breast cancer and irradiation of the internal mammary lymph nodes and does not appear to have a threshold. Lowering heart dose can be achieved by improved planning methods as well as increasing the distance between the target volume and the heart. A deep inspiration breath-hold (DIBH) is often used to this end.

An unassisted DIBH is between 12 and 30 seconds; a simple breast irradiation averages 4 DIBHS for completion. More advanced radiotherapy plans (including lymph nodes) needs up to 20 DIBHs. This great amount is both physically and mentally exhausting.

A protocol was developed to increase breath-hold time using (voluntary) hyperventilation and oxygenation to achieve DIBH times around 3 minutes.

Multiple non-medical interventions are being investigated to prolong a L-DIBH that are feasible in clinical practice. One of these methods will be to alter the time perception of the subjects. It has been noted in multiple studies (both medical and not) that slowing a person's perception of time results in an increase in breath-hold time. This alteration in time perception can be achieved with the use of a slowed clock as well as the usage of mental or physical exercises to preoccupy the subjects.

Other important factors on the duration of breath holds are stress and anxiety, which may also be influenced by (relaxation) exercises (including Abdominal breathing).

The standard protocol for the first phase will be based on the results of the original HOBBIT trial.

40 Volunteers will be asked to perform 3 L-DIBHs each preceded by 3 minutes of hyperventilation at 16 breaths/min with 40L/min at FiO2 60%.

Volunteers will then be randomised into either the standard arm or the intervention arm. The intervention arm will follow standard protocol regarding DIBH preparation, though during the L-DIBH they will be asked to perform a simple mental exercise on a tablet.

Data regarding L-DIBH time, side-effects and volunteer reported stress and comfort will be reported.

Volunteers in each group will be asked to perform 2 series of 3 L-DIBHs on 2 separate days. After having finished these 2 series, there will be a cross-over to the other arm. This cross-over will evaluate the known effect of the learning bias that we see with breath-hold and show whether this effect has an impact on the anticipated benefit of the intervention. With the cross-over we can also ascertain volunteer comfort and preference with each the technique.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer
* Karnofsky index of at least 90
* Able to perform a single DIBH of at least twenty seconds without assistance
* Age ≥ 18 years
* Informed consent obtained, signed and dated before specific protocol procedures
* Female

Exclusion Criteria:

* Pregnant women
* Volunteers above WHO Obesity class II (BMI>35kg/m²)
* Subjects on oxygen treatment during day or night
* COPD or Asthma patients
* Volunteers with pulmonary hypertension
* Gastric tube present
* Smoking
* Previous and substantial breath-holding experience in the past year (e.g., diver, etc.)
* Mental condition rendering the volunteer unable to understand the nature, scope and possible consequences of the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-11-27 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Difference in average L-DIBH time between standard and experimental L-DIBH | 1 year
  Difference in average L-DIBH time between standard and experimental L-DIBH

SECONDARY OUTCOMES:
Patient reported comfort | 1 year
  Comfort on a scale of 0 to 10 where 0 is not comfortable at all and 10 is very comfortable
Patient preferece for standard or experimental L-DIBH setup | 1 year
  What setup do patients prefer
Average L-DIBH time | 1 year
  average time of a L-DIBH (in standard and experimental setup)
Median L-DIBH time | 1 year
  Median time of a L-DIBH (in standard and experimental setup)
Minimum and Maximum L-DIBH time | 1 year
  Minimum and Maximum time of a L-DIBH (in standard and experimental setup)
Oxygen Saturation | 1 year
  Oxygen Saturation during the L-DIBH
Heart Rate | 1 year
  Heart Rate during the hyperventilation and during the L-DIBH
Patient report Pain | 1 year
  Pain on a scale of 0 to 10 where 0 is no pain and 10 is the worst pain possible
Correctness of the mental exercise | 1 year
  A grading (perfect-good-fair-poor) regarding the score achieved during the mental exercise

OTHER OUTCOMES:
Breath-Hold related side-effects | 1 year
  Various side-effects (regarding, nausea, dizziness, coughing, palpitations, cramps)

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital - Radiotherapy Department, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Early Breast Cancer Trialists' Collaborative Group (EBCTCG); Darby S, McGale P, Correa C, Taylor C, Arriagada R, Clarke M, Cutter D, Davies C, Ewertz M, Godwin J, Gray R, Pierce L, Whelan T, Wang Y, Peto R. Effect of radiotherapy after breast-conserving surgery on 10-year recurrence and 15-year breast cancer death: meta-analysis of individual patient data for 10,801 women in 17 randomised trials. Lancet. 2011 Nov 12;378(9804):1707-16. doi: 10.1016/S0140-6736(11)61629-2. Epub 2011 Oct 19. PMID 22019144
- [Background] Darby SC, Ewertz M, McGale P, Bennet AM, Blom-Goldman U, Bronnum D, Correa C, Cutter D, Gagliardi G, Gigante B, Jensen MB, Nisbet A, Peto R, Rahimi K, Taylor C, Hall P. Risk of ischemic heart disease in women after radiotherapy for breast cancer. N Engl J Med. 2013 Mar 14;368(11):987-98. doi: 10.1056/NEJMoa1209825. PMID 23484825
- [Background] Vakaet V, Van Hulle H, Schoepen M, Van Caelenberg E, Van Greveling A, Holvoet J, Monten C, De Baerdemaeker L, De Neve W, Coppens M, Veldeman L. Prolonging deep inspiration breath-hold time to 3 min during radiotherapy, a simple solution. Clin Transl Radiat Oncol. 2021 Feb 23;28:10-16. doi: 10.1016/j.ctro.2021.02.007. eCollection 2021 May. PMID 33732910
- [Background] Schwarz MA, Winkler I, Sedlmeier P. The heart beat does not make us tick: the impacts of heart rate and arousal on time perception. Atten Percept Psychophys. 2013 Jan;75(1):182-93. doi: 10.3758/s13414-012-0387-8. PMID 23143915
- [Background] Vigran HJ, Kapral AG, Tytell ED, Kao MH. Manipulating the perception of time affects voluntary breath-holding duration. Physiol Rep. 2019 Dec;7(23):e14309. doi: 10.14814/phy2.14309. PMID 31833235